CLINICAL TRIAL: NCT04832425
Title: A Phase 2/3 Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of PRAX-114 in Participants With Major Depressive Disorder
Brief Title: A Clinical Trial of PRAX-114 in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAX-114-213
Record Dates: First submitted 2021-03-19; First posted 2021-04-05 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Major Depressive Disorder
Keywords: Mood Disorders; Depressive Disorder; Depression; Depressive Disorder, Unipolar; Depressive Symptoms; Agents, GABA; Receptors, GABA-A; Allosteric Regulation
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRAX-114 (Experimental): 40 mg PRAX-114 once daily
  Interventions: Drug: PRAX-114
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRAX-114 — 40 mg once daily
  Arms: PRAX-114
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial to assess the efficacy and safety of PRAX-114 in participants with moderate to severe major depressive disorder (MDD). Participants will be randomized to receive 28 days of either 40 mg PRAX-114 or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent MDD diagnosis with a current episode duration of at least 8 weeks and no more than 24 months.
2. HAM-D17 total score of ≥23 at Screening and Baseline.
3. Body mass index (BMI) between 18 and 38 kg/m2 (inclusive).

Exclusion Criteria:

1. Lifetime history of seizures, including febrile seizures.
2. Neurodegenerative disorder (eg, Alzheimer's disease, Parkinson's disease, multiple sclerosis, or Huntington's disease).
3. Lifetime history of bipolar disorder, a psychotic disorder (eg, schizophrenia or schizoaffective disorder), or obsessive compulsive disorder or a history of a psychotic mood episode in last 2 years.
4. Any current psychiatric disorder (other than MDD).
5. Lifetime history of treatment resistant depression.
6. Received electroconvulsive therapy (ECT) or vagus nerve stimulation (VNS) within the last year or transcranial magnetic stimulation (TMS) within the last 6 months prior to Screening.
7. Daily consumption of more than 2 standard alcohol-containing beverages for males or more than 1 standard alcohol-containing beverages for females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 17-Item Hamilton Depression Rating Scale (HAM-D17) total score at Day 15 | 15 days
  The HAM-D17 is a depression rating scale consisting of 17 items; 9 items are scored on a 5-point scale (ranging from 0 to 4), and 8 items are scored on a 3-point scale (ranging from 0 to 2). The total score of the 17 items ranges from 0 to 52 with higher scores indicating greater depression. Therefore, a decrease in the total score or on individual item scores indicates improvement.

SECONDARY OUTCOMES:
Change from baseline in HAM-D17 total score at Day 29 | 29 days
  The HAM-D17 is a depression rating scale consisting of 17 items; 9 items are scored on a 5-point scale (ranging from 0 to 4), and 8 items are scored on a 3-point scale (ranging from 0 to 2). The total score of the 17 items ranges from 0 to 52 with higher scores indicating greater depression. Therefore, a decrease in the total score or on individual item scores indicates improvement.
Change from baseline in HAM-D17 total score at all other time points | 8 days, 22 days, 36 days, and 43 days
  The HAM-D17 is a depression rating scale consisting of 17 items; 9 items are scored on a 5-point scale (ranging from 0 to 4), and 8 items are scored on a 3-point scale (ranging from 0 to 2). The total score of the 17 items ranges from 0 to 52 with higher scores indicating greater depression. Therefore, a decrease in the total score or on individual item scores indicates improvement.
Change from baseline in Clinical Global Impression-Severity (CGI-S) score at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The CGI-S assesses the clinician's impression of the participant's current depression symptoms. The clinician should use his/her total clinical experience with this patient population and rate the current severity of the participant's mental illness on a 7-point scale from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients).
Clinical Global Impression-Improvement (CGI-I) score at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to Baseline (Day 1) on a 7-point scale from 1 (Very much improved) to 7 (Very much worse).
HAM-D17 response (reduction from baseline score of ≥50%) at Day 15, Day 29, and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The HAM-D17 is a depression rating scale consisting of 17 items; 9 items are scored on a 5-point scale (ranging from 0 to 4), and 8 items are scored on a 3-point scale (ranging from 0 to 2). The total score of the 17 items ranges from 0 to 52 with higher scores indicating greater depression. Therefore, a decrease in the total score or on individual item scores indicates improvement.
HAM-D17 remission (total score of ≤7) at Day 15, Day 29, and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The HAM-D17 is a depression rating scale consisting of 17 items; 9 items are scored on a 5-point scale (ranging from 0 to 4), and 8 items are scored on a 3-point scale (ranging from 0 to 2). The total score of the 17 items ranges from 0 to 52 with higher scores indicating greater depression. Therefore, a decrease in the total score or on individual item scores indicates improvement.
Change from baseline in the Symptoms of Depression Questionnaire (SDQ) total and sub-scale scores at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The SDQ is a 44-item, self-report scale assessing the severity of symptoms across several subtypes of depression. Items are scored on a 7-point scale (ranging from 1 to 6). The SDQ total score is the sum of all 44 item scores and ranges from 44 to 264 with higher scores indicating worse symptoms.
Patient Global Impression-Improvement (PGI-I) score at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The PGI-I scale is a global self-assessment used to rate the response of a participant's condition to therapy or intervention. It consists of 1 question that asks the participant to rate their current condition compared to how it was prior to beginning treatment on a scale of 1 (very much better) to 7 (very much worse).
Change from baseline in the Work and Social Adjustment Scale (WSAS) at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The WSAS assesses the degree to which mental health problems interfere with day-to-day functioning in 5 domains: work, social leisure activities, private leisure activities, home- management, and personal relationships. The WSAS total score is the sum of the 5 item scores and ranges from 0 to 40, with higher scores indicating poorer adjustment.
Change from baseline in the 12-Item Short Form Survey (SF-12) at Day 15 and all other time points | 8 days, 15 days, 22 days, 29 days, 36 days, and 43 days
  The SF-12 is composed of 12 questions covering 8 dimensions of health: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health. Total scores range from 0 (worse health) to 100 (better health).
Incidence and severity of Adverse Events (AE) | 43 days
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
Incidence of AEs by preferred term | Up to 43 days
  The incidence of AEs will be reported by preferred term, including any terms related to clinically significant changes in body temperature, pulse rate, respiratory rate, blood pressure (systolic and diastolic), clinical laboratory measures (chemistry, hematology, urinalysis, and coagulation), and electrocardiogram parameters (heart rate, PR, QRS, QT, and corrected QT intervals).
Incidence of Columbia-Suicide Severity Rating Scale (C-SSRS) measured suicidal ideation or behavior | Up to 43 days
  The C-SSRS is composed of 5 yes/no questions addressing suicidal behavior and 5 yes/no questions addressing suicidal ideation, with sub-questions assessing the severity. Incidence is measured as the number of "yes" answers indicating the presence of suicidal ideation or behavior.

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Development, Study Director — Praxis Precision Medicines
Locations (31):
- United States (30):
  - Praxis Research Site, Phoenix, Arizona
  - Praxis Research Site, Garden Grove, California
  - Praxis Research Site, Lafayette, California
  - Praxis Research Site, Lemon Grove, California
  - Praxis Research Site, Oceanside, California
  - Praxis Research Site, Pico Rivera, California
  - Praxis Research Site, Redlands, California
  - Praxis Research Site, Jacksonville, Florida
  - Praxis Research Site, Orange City, Florida
  - Praxis Research Site, Orlando, Florida
  - Praxis Research Site, Atlanta, Georgia
  - Praxis Research Site, Decatur, Georgia
  - Praxis Research Site, Chicago, Illinois
  - Praxis Research Site, Gaithersburg, Maryland
  - Praxis Research Site, Worcester, Massachusetts
  - Praxis Research Site, O'Fallon, Missouri
  - Praxis Research Site, Las Vegas, Nevada
  - Praxis Research Site, Berlin, New Jersey
  - Praxis Research Site, Marlton, New Jersey
  - Praxis Research Site, Cedarhurst, New York
  - Praxis Research Site, Rochester, New York
  - Praxis Research Site, Staten Island, New York
  - Praxis Research Site, Dayton, Ohio
  - Praxis Research Site, Allentown, Pennsylvania
  - Praxis Research Site, Media, Pennsylvania
  - Praxis Research Site, Memphis, Tennessee
  - Praxis Research Site, Austin, Texas
  - Praxis Research Site, San Antonio, Texas
  - Praxis Research Site, Charlottesville, Virginia
  - Praxis Research Site, Everett, Washington
- Praxis Research Site, Noble Park, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No